CLINICAL TRIAL: NCT04797845
Title: "Patient's TeleMonitoring With Amyotrophic Lateral Sclerosis Treated by Non Invasive Ventilation at Home." Tele Monitoring Ventilation At Home (TM-VAH)
Brief Title: Patient's TeleMonitoring With Amyotrophic Lateral Sclerosis Treated by Non Invasive Ventilation at Home.
Acronym: TS-VAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0477
Record Dates: First submitted 2021-02-03; First posted 2021-03-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Amyotrophic Lateral Sclerosis; Noninvasive Ventilation
Keywords: Telemonitoring; amyotrophic lateral sclerosis; noninvasive ventilation; feasibility
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- telemonitoring of non invasive ventilation at home (Experimental): Patients will benefit from a quarterly teleconsultation to assess the study criteria through different questionnaires during 12 months. Ventilation machines make it possible to carry out remote monitoring, with the help of healthcare providers.
  Interventions: Other: teleconsultation

INTERVENTIONS:
Other: teleconsultation — Patients will benefit from a quarterly teleconsultation to assess the study criteria through different questionnaires during 12 months.

SUMMARY:
Single-center, prospective pilot study on patients with amyotrophic lateral sclerosis fitted with noninvasive ventilation. The objective is to assess the satisfaction of remote monitoring of patients on non-invasive ventilation after 12 months.

DETAILED DESCRIPTION:
The non invasive ventilation is one of treatments used during the amyotrophic lateral sclerosis when patients have a chronic respiratory failure with alveolar hypoventilation signs. It is demonstrated to improve quality of life and prognosis of the disease. These patients, often severely disabled, generally have a negative experience of repeated hospitalizations. Despite everything, medical and paramedical monitoring is necessary, especially when they are fitted with non invasive ventilation (NIV). A quarterly reassessment is recommended . The possibilities of telemonitoring at home have grown considerably in recent years. In addition, the fans are currently able to remotely transfer a certain amount of data to the service provider, making remote monitoring feasible.Our project therefore aims to assess the feasibility of remote monitoring of patients with Amyotrophic Lateral Sclerosis (ALS) fitted with non invasive ventilation (NIV) through the assessment of their satisfaction, using both medical data and data provided by the ventilator. It is a single-center, prospective pilot study on 30 patients with amyotrophic lateral sclerosis fitted with noninvasive ventilation. Patients will benefit from a quarterly teleconsultation to assess the study criteria through questionnaires during 12 months. Ventilation machines make it possible to carry out remote monitoring, with the help of healthcare providers.

ELIGIBILITY:
o inclusion criteria:

* Patient over 18 years,
* Patient with Amyotrophic Lateral Sclerosis (ALS),
* Already fitted by Non Invasive Ventilation (NIV),
* Patient having signed the informed consent
* Patient affiliated to a social security scheme,
* Patient with a correct understanding of the French language,
* Patient with access to an internet connection at home.

For the caregiver:

* Adult person
* Be the patient's primary caregiver
* Have signed the informed consent intended for the caregiver

  o exclusion criteria:
* Patient with another cause of chronic respiratory failure: other neuromuscular diseases, Chronic obstructive pulmonary disease (COPD), diffuse interstitial lung disease,
* Patient under guardianship or under judicial protection,
* Patient dependent at least 20 hours out of 24 of the non invasive Ventilation (NIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction of the telemonitoring of non invasive ventilation at home assessed by CSQ-8 at the end of the study | 1 year
  Consumer satisfaction questionnaire (CSQ-8), minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.

SECONDARY OUTCOMES:
Effect of remote monitoring | every 3 months during 1 year
  evaluated by teleconsultation
Patient satisfaction during the study | every 3 months during 1 year
  assessed by Consumer satisfaction questionnaire (CSQ-8), minimal score is 8 and maximal score is 32. The best score is 32, that mean that patient is satisfied.
Feasibility for caregivers assessed by Zarit questionnaire | every 3 months during 1 year
  Painfulness or burden assessment scale. Minimal score is 0 and maximal score is 76. the higher the score, the greater the difficulty.
Feasibility for caregivers assessed by Depression Anxiety Stress Scales (DASS-21) questionnaire | every 3 months during 1 year
  Painfulness or burden assessment scale. Minimal score is 0 and maximal score is 63. the higher the score, the greater the depression.
Feasibility for nursing staff | every 3 months during 1 year
  data collected through remote monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Pontier-Marchandise, MD, Principal Investigator — University Hopsital Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No